CLINICAL TRIAL: NCT01807273
Title: Quantification of Biomechanical Parameters of Functional Task Time Up and Go in Hemiplegic Patients
Brief Title: Time Up and go in Hemiplegic Patients
Acronym: TUG
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, Nicolas ROCHE, MDPHD, Centre d'Investigation Clinique et Technologique 805
Other Study IDs: 2012-A01619-3
Record Dates: First submitted 2013-03-07; First posted 2013-03-08 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Difficulty Walking
Keywords: hemiplegic; time up and go test; motion analysis; center of mass
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemiplegic subjects: 60 hemiplegic outpatients walking test
  Interventions: Other: Walking test

INTERVENTIONS:
Other: Walking test
  Other Names: The TUG test included stand up ,walk,turn around ,sit down

SUMMARY:
Investing the Timed Up and Go (TUG) Test in Hemiplegic Patients Using 3D Motion Analysis

DETAILED DESCRIPTION:
The timed up and go is a routine quick test assessing motor functional tasks including stand up ,walk 3 m,turn around and sitting down.We will included hemiplegic patients to quantify biomechanic parameters

ELIGIBILITY:
Inclusion Criteria:

* Patients performing 3D gait analysis
* Male or female adults aged ≥ 18 years,
* Hemiplegia following unique stroke- Patients with hemiplegia able to stand up alone,walk and turn around alone without assistance.

Exclusion Criteria:

* Patient with a protective measure,
* Pregnant women, breastfeeding
* Brain damage bilateral cerebellar syndrome, apraxia and / or severe aphasia,
* Patient who received botulinum toxin injection in the 3 months prior to inclusion, patients who underwent surgery of the locomotor system in the 6 months prior to inclusion,
* No affiliation to a social security
* other pathology, complications with significant impact on the activities of walking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 hemiplegic out patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Variability of the center of mass | 1 hour
  subjects will perform the TUG test with 3D walk analysis equipment

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas ROCHE, MDPHD, Principal Investigator — HOPITAL RAYMOND POINCARE
Locations (1):
- Hopital Raymond Poincare, Garches, Garches, France